CLINICAL TRIAL: NCT05421117
Title: Comparison of Laparoscopic Adnexal Mass Extraction Via the Transumbilical and Transvaginal Routes
Status: Completed | Type: Observational
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, Medical Doctor, associate professor, Erzincan Military Hospital
Other Study IDs: MUGLA-7
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- transumbilical (TU) routes: For the TU group, a surgical glove was created bag during the operation as follows: a sterile, surgical latex glove (size 8.5) was double tied at the level of the wrist, the fingers were removed, and a 75-cm purse-string suture was made using a symmetrical knot to form a bag. The glove bag took an average of 10 min to make. It was lubricated with normal saline to remove the talcum powder and then introduced through the 10-mm umbilical port (optic port). The fingers of the glove were removed to facilitate its insertion with the 10-mm trocar and for ease of movement in the abdominal cavity.
  Interventions: Procedure: Laparoscopic adnexal mass extraction
- transvaginal (TV) routes: A curette was placed into the uterine cavity and stabilized with a tenaculum for manipulation of the uterus. After separation of the adnexal mass ligaments, the manipulator was removed to perform TV retrieval. A vaginal retractor was inserted into the vagina to view the cervix and allow removal of the mass via the TV route. The posterior lip of the cervix was grasped with an Allis forceps and then pulled superiorly to expose the posterior vaginal dome. The sampler was inserted into the vagina and pushed gently against the vaginal wall to define the posterior fornix between the uterosacral ligaments. A 1-2-cm transverse TV posterior colpotomy was performed under laparoscopic control using a 3-mm monopolar hook. The sample was pulled into the vagina by holding the bag mouth from the colpotomy with ring forceps. The bag mouth was opened in the vaginal canal and the sample was transferred from the vagina.

INTERVENTIONS:
Procedure: Laparoscopic adnexal mass extraction — Compared with open procedures, Minimally invasive surgery (MIS) is associated with faster recovery times, better patient quality of life, and lower postoperative complication rates. The removal of an adnexal mass from the abdominal cavity is performed most commonly using the suprapubic, trans umbilical (TU), or trans vaginal (TV) route.
  Groups: transumbilical (TU) routes

SUMMARY:
Adnexal masses are a common clinical problem encountered in gynecological practice. Minimally invasive surgery (MIS) for ovarian pathologies has been adopted widely. Its goals are to minimize abdominal incisions and postoperative pain and to prevent incisional complications, such as incisional hernias and adhesions. Compared with open procedures, MIS is associated with faster recovery times, better patient quality of life, and lower postoperative complication rates. The removal of an adnexal mass from the abdominal cavity is performed most commonly using the suprapubic, umbilical, or vaginal route. Apart from these, mini laparoscopy can provide a better cosmetic result without additional operative time or complications. Despite the limited use of mini laparoscopy for gynecological procedures, its use has increased recently.

After excision, an adnexal mass can be removed through a laparoscopic (LS) port using a variety of endoscopic or containment bags. After the mass has been placed in it, the bag is withdrawn, closed, and expelled through the skin incision with simultaneous trocar removal. When a mass is large or cannot be removed through the port, the incision may be enlarged slightly. This situation may yield a cosmetically worse outcome and increases the risk of postoperative complications, such as adhesion, hernia, and increased postoperative pain. Thus, natural orifice surgery (NOS) has emerged for tissue removal in such cases.

This study was performed to compare the transumbilical (TU) and transvaginal (TV) routes for adnexal mass removal from the abdominal cavity

ELIGIBILITY:
Inclusion Criteria:

-Women who underwent laparoscopic surgery for the removal of benign adnexal masses

Exclusion Criteria:

-Patients with missing data about surgery information

Ages: 16 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women who underwent laparoscopic surgery for the removal of benign adnexal masses at three centers between January 2016 and December 2020 were examined retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incisional pain score | The time between the end of the surgery and 3 hours after the operation
  Each patient was asked by the care nurse or assistant doctor to record the severity of incisional pain on a Visual Analogue Scale (0, no pain; 10, unbearable pain) 3 hours after surgery.

IPD SHARING:
Plan to Share IPD: Undecided